CLINICAL TRIAL: NCT06617104
Title: Explore the Differences in Autonomic Nervous System and Meridian Energy Between Patients With Schizophrenia and Healthy Individuals
Brief Title: Autonomic Nervous System and Meridian Energy in Patients With Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202407147RINC
Record Dates: First submitted 2024-09-02; First posted 2024-09-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Healthy Individuals
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- schizophrenia: According to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), individuals who meet the criteria for a diagnosis of schizophrenia.
  Interventions: Other: no intervention
- healthy individuals: No history of chronic illness in the past and no acute symptoms within the past month.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to explore the differences in autonomic nervous function and meridian energy between schizophrenia patients and healthy individuals. By understanding the meridian and organ conditions of individuals, the study aims to align with the traditional Chinese medicine (TCM) concept of "treating disease before it arises" and provide comprehensive care to patients, thereby improving the quality of care.

DETAILED DESCRIPTION:
Data collection was conducted at a medical center in northern Taiwan. Sample size estimation was performed using G*Power 3.1. A total of 50 patients with schizophrenia were assigned to the disease group, and 50 healthy individuals were assigned to the control group, with a total of 100 participants expected. Data collection included: personal demographic questionnaire, body constitution questionnaire (BCQ), WHOQOL-BREF (Taiwan version) for quality of life, brief psychiatric rating scale (BPRS), heart rate variability (HRV), meridian energy

ELIGIBILITY:
Inclusion Criteria:

1. Disease group：

   * Diagnosed with schizophrenia by a physician (ICD-10 code F20, such as F20.0, F20.1, F20.2, F20.3, F20.5, F20.89, or F20.9), with stable condition, and has not had any changes in medication dosage or admission to a psychiatric acute care unit in the past 3 months.
   * Aged between 18 and 65 years.
   * Able to understand, speak, read, and write Mandarin or Taiwanese.
2. Control group：

   * No history of chronic illness and no acute symptoms within the past month.
   * Aged between 18 and 65 years.
   * Able to understand, speak, read, and write Mandarin or Taiwanese.

Exclusion Criteria:

1. Disease group：

   * Individuals with cardiovascular conditions, severe neurological disorders (e.g., organic brain disorders, early-stage dementia or diagnosed dementia), or substance abuse issues.
   * Individuals who have used medications affecting the autonomic nervous system within the past month, such as mood stabilizers, antidepressants, angiotensin-converting enzyme inhibitors inhibitors, β-blockers, or antiarrhythmics.
   * Individuals with metallic implants that could affect heart rate variability.
   * Individuals with involuntary and uncontrollable body tremors.
   * Women currently menstruating.
   * Pregnant women.
2. Control group：

   * Individuals with cardiovascular conditions, severe neurological disorders (e.g., organic brain disorders, early-stage dementia or diagnosed dementia), or substance abuse issues.
   * Individuals who have used medications affecting the autonomic nervous system within the past month, such as psychiatric medications, angiotensin-converting enzyme inhibitors inhibitors, β-blockers, or antiarrhythmics .
   * Individuals with metallic implants that could affect heart rate variability.
   * Individuals with involuntary and uncontrollable body tremors.
   * Women currently menstruating.
   * Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Disease group(schizophrenia):According to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), individuals who meet the criteria for a diagnosis of schizophrenia.
  2. Control group(healthy individuals):No history of chronic illness in the past and no acute symptoms within the past month.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2025-08-19 (Estimated)

PRIMARY OUTCOMES:
meridian energy | This study is a cross-sectional study with a single follow-up. Participants who meet the inclusion criteria will be included in the study, with a recruitment period of one year.
  Measuring the body energy under static balance conditions using principles of electromagnetic induction technology.The measurement items include:lung meridian (LU), large intestine meridian (LI), stomach meridian (ST), spleen meridian (SP), heart meridian (HT), small intestine meridian (SI), bladder meridian (BL), kidney meridian (KI), pericardium meridian (PC), triple burner meridian (SJ), gallbladder meridian (GB), liver meridian (LR)
heart rate variability | This study is a cross-sectional study with a single follow-up. Participants who meet the inclusion criteria will be included in the study, with a recruitment period of one year.
  Assessing autonomic nervous system activity through the measurement of RR intervals. The measurement items include: the square root of the mean squared differences of successive NN intervals , NN50 count divided by the total number of all NN intervals, HRV triangular index, low frequency power, high frequency power, LF/HF Ratio, total power

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No